CLINICAL TRIAL: NCT00466401
Title: Phase 4 Study on Effect of Ezetimibe on Platelet Aggregation and LDL Tendency to Peroxidation In Hypercholesterolemic Patients on Simvastatin
Brief Title: Effect of Ezetimibe on Platelet Aggregation and LDL Tendency to Peroxidation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-5-155-S
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin; Ezetimibe

INTERVENTIONS:
Drug: Simvastatin
Drug: Ezetimibe

SUMMARY:
The aim of our study is to Estimate the reduction of LDL by ezetimibe in hypercholesterolemic patients on simvastatin.Investigate the effect of LDL lowering by ezetimibe on platelet activity and LDL tendency to peroxidation in hypercholesterolemic patients on simvastatin therapy

The hypothesis is that:

1. LDL lowering by ezetimibe on-top of simvastatin in patients on fixed dose of simvastatin can reduce platelet aggregation, due to the potential decreasing of cholesterol content in the platelet membranes.
2. LDL lowering by ezetimibe can lower LDL tendency to peroxidation.

ELIGIBILITY:
Inclusion Criteria:

1. Hypercholesterolemic patients on stable simvastatin dose for at least one month.
2. Age ≥18 years on stable AHA step 1 diet.
3. Patients without CHD or with one risk factors ; LDL > 130 mg/dL and for Patients with CHD or CHD risk equivalent(clinical manifestations of non-coronary forms of atherosclerotic disease) or with 2 risk f actors (cigarette smoking, hypertension (BP ≥140/90 mm Hg or on antihypertensive medication), low HDL cholesterol (<40 mg/dL), family history of premature CHD;LDL>100 mg/dL
4. Patients 'on at least simvastatin treatment of 20 mg per day.
5. CPK, ALT and AST < 1.5 X upper limit of normal at baseline.

Exclusion Criteria:

1. Women currently receiving cyclical hormones.
2. Treatment with psyllium, other fiber based laxatives, phytosterol margarines, or other OTCs that affect serum lipids, unless treated with a stable regimen for > 6 weeks and the patient agrees to continue this regimen for the duration of the trial.
3. Oral corticosteroids unless used as replacement therapy for pituitary/adrenal disease and a stable regimen for at least 6 weeks.
4. Lipid lowering agents including fish oils and QUESTRAN taken within 6 weeks.
5. Active coronary heart disease: unstable angina, acute myocardial infarction, CABG or PTCA within the last 3 months.
6. Women with childbearing potential unless on safe contraception.
7. Psychiatric disease with defect in judgement.
8. Severe renal or hepatic disease.
9. Uncontrolled hypo- or hyperthyroidism.
10. Contraindication for ezetimibe or simvastatin treatment. The patients will continue on their treatment with simvastatin for 6 weeks, and then the patients will be treated by the same dose of simvastatin combined with ezetimibe 10 mg/day for other 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamah Hussein, MD, Principal Investigator — Ziv Hospital
Locations (1):
- Internal Medicine Department A ,Ziv Goverment Hospital, Safed, Israel

REFERENCES:
- [Background] Bays HE, Moore PB, Drehobl MA, Rosenblatt S, Toth PD, Dujovne CA, Knopp RH, Lipka LJ, Lebeaut AP, Yang B, Mellars LE, Cuffie-Jackson C, Veltri EP; Ezetimibe Study Group. Effectiveness and tolerability of ezetimibe in patients with primary hypercholesterolemia: pooled analysis of two phase II studies. Clin Ther. 2001 Aug;23(8):1209-30. doi: 10.1016/s0149-2918(01)80102-8. PMID 11558859
- [Background] Davidson MH, McGarry T, Bettis R, Melani L, Lipka LJ, LeBeaut AP, Suresh R, Sun S, Veltri EP. Ezetimibe coadministered with simvastatin in patients with primary hypercholesterolemia. J Am Coll Cardiol. 2002 Dec 18;40(12):2125-34. doi: 10.1016/s0735-1097(02)02610-4. PMID 12505224
- [Background] van Heek M, Austin TM, Farley C, Cook JA, Tetzloff GG, Davis HR. Ezetimibe, a potent cholesterol absorption inhibitor, normalizes combined dyslipidemia in obese hyperinsulinemic hamsters. Diabetes. 2001 Jun;50(6):1330-5. doi: 10.2337/diabetes.50.6.1330. PMID 11375333
- [Background] Sager PT, Melani L, Lipka L, Strony J, Yang B, Suresh R, Veltri E; Ezetimibe Study Group. Effect of coadministration of ezetimibe and simvastatin on high-sensitivity C-reactive protein. Am J Cardiol. 2003 Dec 15;92(12):1414-8. doi: 10.1016/j.amjcard.2003.08.048. PMID 14675576
- [Background] Davis HR Jr, Compton DS, Hoos L, Tetzloff G. Ezetimibe, a potent cholesterol absorption inhibitor, inhibits the development of atherosclerosis in ApoE knockout mice. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):2032-8. doi: 10.1161/hq1201.100260. PMID 11742881
- [Background] Lavy A, Brook GJ, Dankner G, Ben Amotz A, Aviram M. Enhanced in vitro oxidation of plasma lipoproteins derived from hypercholesterolemic patients. Metabolism. 1991 Aug;40(8):794-9. doi: 10.1016/0026-0495(91)90005-h. PMID 1861629
- [Background] Hussein O, Frydman G, Frim H, Aviram M. Reduced susceptibility of low density lipoprotein to lipid peroxidation after cholestyramine treatment in heterozygous familial hypercholesterolemic children. Pathophysiology. 2001 Aug;8(1):21-28. doi: 10.1016/s0928-4680(01)00061-x. PMID 11476969
- [Background] Surya II, Akkerman JW. The influence of lipoproteins on blood platelets. Am Heart J. 1993 Jan;125(1):272-5. doi: 10.1016/0002-8703(93)90096-r. No abstract available. PMID 8380241
- [Background] Ardlie NG, Selley ML, Simons LA. Platelet activation by oxidatively modified low density lipoproteins. Atherosclerosis. 1989 Apr;76(2-3):117-24. doi: 10.1016/0021-9150(89)90094-4. PMID 2730708
- [Background] Osamah H, Mira R, Sorina S, Shlomo K, Michael A. Reduced platelet aggregation after fluvastatin therapy is associated with altered platelet lipid composition and drug binding to the platelets. Br J Clin Pharmacol. 1997 Jul;44(1):77-83. doi: 10.1046/j.1365-2125.1997.00625.x. PMID 9241100
- [Background] Aviram M. Plasma lipoprotein separation by discontinuous density gradient ultracentrifugation in hyperlipoproteinemic patients. Biochem Med. 1983 Aug;30(1):111-8. doi: 10.1016/0006-2944(83)90013-3. PMID 6626183
- [Background] Knopp RH, Gitter H, Truitt T, Bays H, Manion CV, Lipka LJ, LeBeaut AP, Suresh R, Yang B, Veltri EP; Ezetimibe Study Group. Effects of ezetimibe, a new cholesterol absorption inhibitor, on plasma lipids in patients with primary hypercholesterolemia. Eur Heart J. 2003 Apr;24(8):729-41. doi: 10.1016/s0195-668x(02)00807-2. PMID 12713767